CLINICAL TRIAL: NCT06213610
Title: Open-label Randomized Crossover Two Period Single Dose Bioequivalence Study of Two Formulations of Perindopril (Perindopril Tert-butylamine) 8 mg (Pharmtechnology LLC, Republic of Belarus) and Prestarium® A 10 mg (Perindopril Arginine) 10 mg Tablets (Les Laboratoires Servier Industrie, France) in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Perindopril Tablets in Healthy Volunteers Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharmtechnology LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BE-PER01-23
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Perindopril

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Other): 25 subjects assigned to the sequence TR will receive a single oral dose of the test product Perindopril 8 mg tablet, marked as T in the sequence, in Period 1 and a single oral dose of the reference product Prestarium® A 10 mg tablet, marked as R in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Perindopril tablet; Drug: Prestarium® A tablet
- Sequence RT (Other): 25 subjects assigned to the sequence RT will receive a single oral dose of the reference product Prestarium® A 10 mg tablet, marked as R in the sequence, in Period 1 and a single oral dose of the test product Perindopril 8 mg tablet, marked as T in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Perindopril tablet; Drug: Prestarium® A tablet

INTERVENTIONS:
Drug: Perindopril tablet — Perindopril is manufactured by Pharmtechnology LLC, Republic of Belarus. Each tablet contains 8 mg of perindopril tert-butylamine.
  Other Names: The test product
Drug: Prestarium® A tablet — Prestarium® A is manufactured by Les Laboratoires Servier Industrie, France. Each tablet contains 10 mg of perindopril arginine.
  Other Names: The reference product

SUMMARY:
This is an open-labeled, randomized, two period, single-center, crossover, comparative study, where each participant will be randomly assigned to the reference (Prestarium ® A 10 mg tablets) or the test (Perindopril 8 mg tablets) formulation in each period of study (sequences Test-Reference (TR) or Reference-Test (RT)), in order to evaluate if both formulations are bioequivalent.

DETAILED DESCRIPTION:
This is an open-labeled, randomized, two period, crossover, a single-center, comparative, single-dose study, in which 50 healthy adult subjects will receive one of the study treatments during each study period.

The objective of this study is to determine the bioequivalence of two different formulations of Perindopril after a single oral dose administration under fasting conditions.

Subject eligibility for this study will be determined at the screening visit and eligible subjects will be admitted to the clinical research unit at least 12 hours prior to drug administration for each study period.

Hospitalization in the first period of the study will last no more than 36 hours, after which, in the absence of indications for an extension of hospitalization, each subject will be released home; after that, the first period of the study will be completed.

The procedures of the second study period will be identical to the first period.

After completing all the procedures of the second study period, each subject will undergo a final examination, after which, in case of the absence of adverse events and indications for prolonging hospitalization, the study for the subjects will be considered completed.

The total duration of the study for the subject will be no more than 60 days.

Eligible subjects will be randomized to one of two treatment sequences. There will be two sequences in the study: TR and RT, where T = the test product, R = the reference product.

For each study period, subjects will receive a single oral dose of perindopril (the test or the reference formulation). Study participants will be aware they will receive different formulations of the same drug, without being informed which product (Test or Reference) is being administered. For each subject, all scheduled postdose activities and assessments will be performed relative to the time of study drug administration.

Fasting will continue for at least 4 hours following drug administration, after which a standardized lunch will be served. Next meals will be provided for subjects in 4 hours, 8 hours and 12 hours after drug administration.

Water will be provided as needed until 1 hour predose. Water will be allowed beginning 2 hours after the administration of the drug.

A total of 28 blood samples will be collected (one tube of 5-10 mL each) in each study period for pharmacokinetic (PK) assessments. The first blood sample will be collected prior to drug administration while the others will be collected up to 72 hours after drug administration.

Perindopril and perindoprilate plasma concentrations will be measured according to a validated bioanalytical method.

Statistical analysis of all PK parameters will be based on an ANOVA model. Two-sided 90% confidence interval of the ratio of geometric LSmeans obtained from the ln-transformed PK parameters will be calculated.

Statistical inference of perindopril and perindoprilate will be based on a bioequivalence approach using the following standards: the ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the Test and the Reference for the ln-transformed parameters Cmax and AUC0-t should all be within the 80.00 to 125.00% bioequivalence range.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy european men or women aged between 18 to 45 years
2. Body mass index 18.5-30 kg/m² according to Quetelet's weight-height index
3. Verified diagnosis "healthy" according to the anamnesis data and the results of standard clinical, laboratory and instrumental examination methods, physical examination and anamnestic examination
4. The level of systolic blood pressure (SBP) measured in the sitting position at the time of screening ≥100 mm Hg and ≤ 139 mm Hg and diastolic blood pressure (DBP) ≥ 60 mm Hg or ≤ 90 mm Hg; heart rate more than 60 beats/min and less than 90 beats/min at the time of screening, respiratory rate more than 12 and less than 20 per minute at the time of screening, body temperature above 35.9 ° C and below 36.9 °C at the time of screening
5. Subjects are able to understand the requirements of the study
6. Subjects are able to accept all the restrictions imposed during the course of the study
7. The written consent of the volunteer to be included in the study
8. For female subject:

   * negative pregnancy test;
   * adherence to reliable methods of contraception for female of childbearing potential: sexual continence, or condom + spermicide, or diaphragm + spermicide, started at least 14 days before the first dose of the study drug; intrauterine contraception is also a reliable method of contraception, installed at least 4 weeks before taking the study drugs in the first period;
   * сonsent to use these methods of contraception within 30 days after taking the drug in the second period;
   * women who do not use acceptable methods of contraception, if they are considered incapable of childbearing, will also be able to participate in the study: women who have undergone a hysterectomy or tubal ligation, women with a clinical diagnosis of infertility, and women who are in menopause (at least a year without menstruation in the absence of alternative pathologies that may cause the cessation of menstruation);
   * in case of using contraceptives (injectable and oral hormonal contraceptives, subcutaneous hormonal implants or intrauterine hormonal therapeutic systems), the latter should be canceled at least 60 days before taking the drug in the first period;
9. For male: consent to use a double barrier method of contraception (condom + spermicide) or complete sexual abstinence, as well as consent not to participate in sperm donation during the entire study and 30 days after taking the drug in the second period.

Exclusion Criteria:

1. hypersensitivity to perindopril or any ACE inhibitors, amlodipine, indapamide or excipients that are part of any of the investigational drugs, or intolerance to these components;
2. burdened allergic history
3. lactose intolerance, lactase deficiency, glucose-galactose malabsorption.
4. acute infectious diseases or allergic diseases that ended less than 4 weeks before taking the drug in the first period;
5. surgical interventions on the gastrointestinal tract, with the exception of appendectomy
6. clinically significant pathologies of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys and blood;
7. the value of standard laboratory and instrumental parameters that go beyond the reference values
8. positive test for syphilis, hepatitis B, hepatitis C or HIV at the time of screening;
9. positive test for alcohol in exhaled air at screening
10. positive urine analysis for the content of narcotic and potent substances during screening (opiates, morphine, barbiturates, benzodiazepines, cannabinoids/marijuana)
11. for women - positive pregnancy test at screening
12. adherence to any low-sodium diet within 2 weeks prior to taking the drug in the first study period, or adherence to a special diet (vegetarian, vegan, salt-restricted)
13. intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of dry wine or 50 ml of spirits ethyl 40%) or history of alcoholism, drug addiction, drug abuse;
14. inability to go without food for at least 12 hours and the inability to take the drug on an empty stomach;
15. donation of plasma or blood (450 ml or more) less than 3 months before taking the drug in the first period;
16. the use of injectable and oral hormonal contraceptives for 60 days before taking the drug in the first period;
17. the use of subcutaneous hormonal implants or intrauterine hormonal therapeutic systems for 6 months before taking the drug in the first period;
18. use of any prescription and OTC drugs less than 2 weeks before the screening
19. use of well-known inducers of liver microsomal enzymes (barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole, etc.) inhibitors of liver microsomal enzymes (antidepressants, cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines), vitamins, herbs and food additives (cat's claw, angelica officinalis, oenothera, pyrethrum, garlic, ginger, ginkgo, red clover, horse chestnut, green tea, ginseng; St. john's wort etc.) less than 30 days before enrollement in the study
20. for women: volunteers with preserved reproductive potential who had unprotected sexual intercourse with an unsterilized male partner within 30 days before the first day of screening;
21. breastfeeding;
22. participation in other clinical trials of drugs less than 3 months before the screening;
23. difficulty with taking blood;
24. smoking
25. volunteers who are unwilling or unable to give up alcohol and excessive physical activity from the first day of screening until the follow-up visit;
26. consumption of caffeine and xanthine-containing drinks and products (tea, coffee, chocolate, cola, etc.), products containing poppy seeds and use of citrus fruits (including grapefruit and grapefruit juice) from the first day of screening until the follow-up visit;
27. intense physical activity or following lifestyle (night work, extreme physical activity)
28. lack of intention of volunteers to comply with the Protocol requirements throughout the course of the study and/or lack, in the opinion of the Investigator, of the volunteers' ability to understand and evaluate the information on this study as part of the informed consent form signing process, in particular regarding the expected risks and possible discomfort;
29. dehydration due to diarrhea, vomiting or other reason within the last 24 hours before taking the drug in the first period of the study;
30. the presence of seizures, epilepsy and any other neurological disorders in the history of volunteers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-03-06 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Cmax of perindopril after administration of the test and the reference products. | Time points for perindopril 0.00 (prior to each drug administration) and 0.05, 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 12.00, 24.00 hours after each drug administration
  Maximum observed concentration in plasma
AUC0-72 of perindopril after administration of the test and the reference products | Time points for perindopril 0.00 (prior to each drug administration) and 0.05, 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 12.00, 24.00 hours after each drug administration
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration (TLQC) using the linear trapezoidal method
Cmax of perindoprilat after administration of the test and the reference products | Time points for perindoprilat 0.00 (prior to each drug administration) and 0.30, 1.00, 1.30, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 5.30, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration
  Maximum observed concentration in plasma
AUC0-72 of perindoprilat after administration of the test and the reference products | Time points for perindoprilat 0.00 (prior to each drug administration) and 0.30, 1.00, 1.30, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 5.30, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00 hours after each drug administration.
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration (TLQC) using the linear trapezoidal method

SECONDARY OUTCOMES:
Tmax of perindopril in plasma after administration of the test and the reference products. | Up to 24 hours
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value
Tmax of perindoprilat in plasma after administration of the test and the reference products. | Up to 72 hours
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value.
AUC0-INF of perindopril in plasma after administration of the test and the reference products. | Up to 24 hours
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-t + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant).
AUC0-INF of perindopril in plasma after administration of the test and the reference products. | Up to 72 hours
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-t + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant).
Terminal elimination half-life (Thalf) of perindopril in plasma after administration of the test and the reference products. | Up to 24 hours
  Terminal elimination half-life, calculated as ln(2)/λZ.
Terminal elimination half-life (Thalf) of perindoprilat in plasma after administration of the test and the reference products. | Up to 72 hours
  Terminal elimination half-life, calculated as ln(2)/λZ.
Number of treatment-emergent adverse events for the test and the reference products. | Up to 60 days
  The safety population will include all subjects who received at least one dose of the test or the reference product. Any significant changes will be recorded as treatment-emergent adverse events only if they are judged clinically significant by the qualified investigator or delegate

CONTACTS AND LOCATIONS:
Locations (1):
- Ligand Research LLC, Moscow, Russia